CLINICAL TRIAL: NCT00599287
Title: Methylphenidate, Rivastigmine or Haloperidol in Hypoactive Delirium in Intensive Care Patients: a Randomized, Mono-blind Pilot Trial
Brief Title: Methylphenidate, Rivastigmine or Haloperidol in Hypoactive Delirium in Intensive Care Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inclusion rate too low due to a lack of eligible patients and difficulties obtaining informed consent.
Sponsor: UMC Utrecht (Other)
Responsible Party: prof. dr. J. Kesecioglu, University Medical Center Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICHYPDEL/002; METC-UMCU 07/236
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2008-02

CONDITIONS: Delirium
Keywords: ICU delirium; Hypoactive delirium; Haloperidol; Methylphenidate; Rivastigmine; Hypoactive ICU delirium
MeSH Terms: conditions — Delirium | interventions — Haloperidol; Methylphenidate; Rivastigmine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): No intervention
- 2 (Experimental): Methylphenidate
  Interventions: Drug: Methylphenidate
- 3 (Experimental): Rivastigmine
  Interventions: Drug: Rivastigmine
- 4 (Experimental): Haloperidol
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Haloperidol — Haloperidol 2,5 mg. 2 dd 1, oral. (if patient is 69 years or younger) Haloperidol 1 mg. 2 dd 1, oral (if patient is 70 years or older)
  Other Names: Haldol
  Arms: 4
Drug: Methylphenidate — Methylphenidate 5 mg. 2 dd 1, oral, increased every day with 10 mg. until negative CAM(-ICU) or side-effects. Maximum dosage 30 mg./day
  Other Names: Ritalin
  Arms: 2
Drug: Rivastigmine — Rivastigmine 1,5 mg. 2 dd 1, oral, increased every third day with 3 mg. until negative CAM(-ICU) or side-effects. Maximum dosage 12 mg./day
  Other Names: Exelon
  Arms: 3

SUMMARY:
The purpose of this pilot-trial is the feasibility of a large randomized, placebo controlled, doubleblind clinical trial to investigate the use of methylphenidate, rivastigmine or haloperidol in hypoactive ICU-delirium. In addition we will compare duration of delirium, severity of delirium, length of ICU/hospital stay and side effects between the different interventions.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Diagnosed as hypoactive delirium
* Informed consent given

Exclusion Criteria:

* Pregnancy
* Epilepsy
* M. Parkinson
* Lewy-body dementia
* Prolonged QT-time
* Known allergy to the medicinals used
* Renal replacement therapy
* Hepatic encephalopathy
* Hyperthyroid
* Glaucoma
* Previous suicide attempts
* Syndrome of Gilles de la Tourette
* Patients which cannot receive the medication oral or through a nasogastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
duration of delirium | Days

SECONDARY OUTCOMES:
duration of ICU-stay | days
duration of in hospital stay | days
delirium severity | duration of delirium
frequency of side effects | duration of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Kesecioglu, MD PhD, Study Director — UMC Utrecht
Locations (1):
- University Medical Center, Utrecht, Netherlands